CLINICAL TRIAL: NCT04529668
Title: Effect of Vitamin d Deficiency in Chronic Rhinosinusitis With Nasal Polyposis: Clinical, Laboratory & Immunohistochemical Study
Brief Title: Effect of Vitamin d Deficiency in Chronic Rhinosinusitis With Nasal Polyposis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammad Salah Mohammad Mahmoud, Doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASUMD241/2015
Record Dates: First submitted 2020-08-25; First posted 2020-08-27 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Vitamin D Deficiency, Nasal Polyposis
Keywords: VITAMIN D DEFICIENCY, CHRONIC RHINOSINUSITIS WITH NASAL POLYPOSIS
MeSH Terms: conditions — Vitamin D Deficiency; Nasal Polyps

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: all will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Experimental): twenty-five patients with the clinical diagnosis of chronic rhinosinusitis with nasal Polyposis will receive vitamin D supplementation
  Interventions: Drug: vitamin D supplementation
- group II (Active Comparator): twenty-five patients with the clinical diagnosis of chronic rhinosinusitis with nasal Polyposis will NOT receive vitamin D supplementation
  Interventions: Drug: usual therapy for nasal polyposis

INTERVENTIONS:
Drug: vitamin D supplementation — vitamin D supplementation
  Arms: group I
Drug: usual therapy for nasal polyposis — steroids ( systemic and local )
  Arms: group II

SUMMARY:
Aim of the work

1. To determine if chronic rhinosinusitis with nasal polyps' (CRSwNP) populations are vitamin D deficient.
2. To determine the possible anti-inflammatory effect of vitamin D supplementation (clinically & histologically). & investigate its relation to immunohistochemical tissue expression of basic fibroblast growth factor

DETAILED DESCRIPTION:
Patients & methods

Study groups:

Fifty patients with the clinical diagnosis of chronic rhinosinusitis with nasal Polyposis (CRSwNP) resistant to medical treatment at Otorhinolaryngology outpatient clinic, Ain Shams University hospitals. Group I : twenty five patients will receive vitamin D supplementation, while group II won't receive vitamin D supplementation.

Inclusion criteria:

Patients (18-60) years of age with clinical diagnosis of chronic rhinosinusitis with nasal Polyposis (CRSwNP) resistant to medical treatment at Otorhinolaryngology outpatient clinic, Ain Shams University hospital.

Both groups (I & II) will be subjected to venous blood sampling and 25(OH) vitamin D level measurement & will be subjected to:

1. Careful history taking.
2. Complete ENT examination and endoscopic evaluation of the nose.
3. CT scan paranasal sinuses coronal and axial view to evaluate the affected sinuses.
4. Vitamin D3 serum level (before Vitamin D3 supplementation).
5. Biopsy from nasal polyps & immunohistochemical assessment (before Vitamin D3 supplementation).
6. Vitamin D3 supplementation 50000 IU/weekly for 6 weeks.
7. Vitamin D3 serum level (after Vitamin D3 supplementation).
8. Biopsy from nasal polyps & immunohistochemical assessment (after Vitamin D3 supplementation).

Exclusion criteria:

* Pregnant and lactating females.
* Patients taking multivitamins containing vitamin D for at least six months.
* Immune deficiency or suppression.
* Ciliary motility disorders.
* Wegner's granulomatosis and other granulomatous diseases.
* Sino-nasal malignancy.

  1. History:

     1. Personal history: name, age, sex, occupation and environment (smoking, exposure to irritants).
     2. Complaint and history of present illness: analysis of the patient's chief complaints with special emphasis on CRS symptoms.
     3. Medical history: Previous medical treatment for CRS (antibiotics, topical and systemic corticosteroids, etc...) or for any other disease (allergy, hypertension, asthma, GERD, etc...) including questions about the dose and duration of treatment and the achieved results. It included also past history of surgery.
     4. Family history: History of allergy, asthma, polyposis, migraine, genetic diseases, etc….
  2. Examination:

     1. General examination: it will be done for all patients as a routine.
     2. Local examination (complete ENT examination): Oral, laryngeal and ear examination will be done to exclude other ENT disease and then careful nasal examination will be done.
     3. Endoscopic examination: Diagnostic nasal endoscopy will be done for all patients.
  3. Investigations:

     A- CT scans will be done (in coronal, axial planes) for all patients with chronic rhinosinusitis with nasal Polyposis (CRSwNP).

     B- 25-OH Vitamin D serum level: (before & after vitamin D supplementation)
  4. Biopsy from nasal polyps :

     Tissue samples will be taken from the nasal polyps of all patients with chronic rhinosinusitis with nasal Polyposis (CRSwNP) at the start of the study (before VD therapy) under local anesthesia at the outpatient clinic for histological (epithelium, basal lamina, lamina propria, cells, blood vessels) & immunohistochemical (basic fibroblast growth factors) examination.
  5. Vitamin D3 supplementation:

     Vitamin D3 (cholecalciferol) will be given to the study group Ia orally 50000 IU weekly for 6 weeks. In addition to local nasal steroids & saline nasal wash. All patients will be monitored by serum calcium level. While group Ib will not be given vitamin D supplementation.
  6. Biopsy from nasal polyps :

Tissue samples will be taken from the nasal polyps of all patients with chronic rhinosinusitis with nasal Polyposis (CRSwNP) after vitamin D supplementation for immunohistochemical assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients (18-60) years of age with clinical diagnosis of chronic rhinosinusitis with nasal Polyposis (CRSwNP) at Otorhinolaryngology outpatient clinic, Ain Shams University hospital.

Exclusion Criteria:

* • Pregnant and lactating females.

  * Patients taking multivitamins containing vitamin D for at least six months.
  * Immune deficiency or suppression.
  * Ciliary motility disorders.
  * Wegner's granulomatosis and other granulomatous diseases.
  * Sino-nasal malignancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-20 (Estimated)

PRIMARY OUTCOMES:
patient complaint | 6 weeks
  by SNOT-22 , Sino-nasal Outcome Test , completion of the SNOT-22 prior to and following Vitamin D supplementation . Each subject completed the SNOT-22 during a clinic visit by answering all questions based on a 0-5 scale, where 0 defines no problems with the given symptom and 5 defines maximal problems
examintaion | 6 weeks
  Lund & Kennedy endoscopic appearance score, examination will be done before and after vitamin D supplementation , with 0 means absent finding and 2 means worst finding
histopathology | 6 weeks
  immunohistochemitsry for fibroblast growth factor

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams Univesrity, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fokkens WJ, Lund VJ, Mullol J, Bachert C, Alobid I, Baroody F, Cohen N, Cervin A, Douglas R, Gevaert P, Georgalas C, Goossens H, Harvey R, Hellings P, Hopkins C, Jones N, Joos G, Kalogjera L, Kern B, Kowalski M, Price D, Riechelmann H, Schlosser R, Senior B, Thomas M, Toskala E, Voegels R, Wang de Y, Wormald PJ. EPOS 2012: European position paper on rhinosinusitis and nasal polyps 2012. A summary for otorhinolaryngologists. Rhinology. 2012 Mar;50(1):1-12. doi: 10.4193/Rhino12.000. PMID 22469599